CLINICAL TRIAL: NCT06842823
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Navenibart in Participants With Hereditary Angioedema (HAE)
Brief Title: A Study of Navenibart in Participants With Hereditary Angioedema
Acronym: ALPHA-ORBIT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astria Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STAR-0215-301
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: HAE; Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema

STUDY DESIGN:
Intervention Model Description: Adult participants will be randomly assigned to one of 4 arms. Adolescent participants will be assigned to a single experimental group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Adult Navenibart Dosing Regimen 1 (Experimental): Participants will receive 600 mg of navenibart every 3 months.
  Interventions: Drug: navenibart
- Adult Navenibart Dosing Regimen 2 (Experimental): Participants will receive 600 mg of navenibart on Day 1 and 300 mg every 3 months starting at month 3.
  Interventions: Drug: navenibart
- Adult Navenibart Dosing Regimen 3 (Experimental): Participants will receive 600 mg of navenibart every 6 months.
  Interventions: Drug: navenibart
- Placebo (adult) (Placebo Comparator): Participants will receive placebo every 3 months.
  Interventions: Drug: Placebo
- Adolescent Navenibart Dosing Regimen 1 (Experimental): Participants will receive 600 mg of navenibart on Day 1 and 300 mg every 3 months starting at month 3.
  Interventions: Drug: navenibart

INTERVENTIONS:
Drug: navenibart — Navenibart will be administered as a subcutaneous injection.
  Other Names: STAR-0215
  Arms: Adolescent Navenibart Dosing Regimen 1; Adult Navenibart Dosing Regimen 1; Adult Navenibart Dosing Regimen 2; Adult Navenibart Dosing Regimen 3
Drug: Placebo — Placebo will be administered as a subcutaneous injection.
  Arms: Placebo (adult)

SUMMARY:
This is a Phase 3 multicenter, randomized, double-blind, placebo-controlled clinical trial evaluating the safety and efficacy of subcutaneous administration of navenibart in adult and adolescent participants with type 1 or type 2 hereditary angioedema (HAE). The goal of this clinical trial is to evaluate the efficacy and safety of navenibart compared to placebo in preventing HAE attacks in participants with HAE.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of HAE (Type 1 or 2). The following must be met:

  1. Documented clinical history consistent with HAE
  2. Lab findings consistent with HAE Type 1 or 2
* Experienced at least 2 HAE attacks during the Run-In period, as confirmed by an investigator based on meeting the protocol-specified definition of an HAE attack.

Exclusion Criteria:

* Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1 inhibitor deficiency, HAE with normal C1-INH (also known as HAE type 3), idiopathic angioedema, or angioedema associated with urticaria.
* Use of therapies prescribed for the prevention of HAE attacks may not be used during the trial or within the below time frames prior to the Run-In Period (adult participants may be on these medications at the time of the Screening Visit, but will need to washout prior to entering the Run-In Period).

  1. Tranexamic acid, oral danazol, oral stanazolol, and oral oxandrolone within 3 days prior to Run-In
  2. Plasma-derived C1INH for LTP within 14 days prior to Run-In
  3. Berotralstat within 21 days prior to Run-In
  4. Lanadelumab within 70 days prior to Run-In
  5. Garadacimab within 90 days prior to Run-In

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of time-normalized investigator-confirmed HAE attacks during the 6-month Treatment Period. | Day 1 through Day 181

SECONDARY OUTCOMES:
Number of moderate or severe investigator-confirmed HAE attacks during the 6-month Treatment Period. | Day 1 through Day 181
Number of investigator-confirmed HAE attacks that require on-demand treatment during the 6-month Treatment Period. | Day 1 through Day 181
Percent reduction in monthly investigator-confirmed HAE attacks in the 6-month Treatment Period versus the Run-In Period. | Baseline through Day 181
Time to first investigator-confirmed HAE attack after first and second dose. | Day 1 through Day 181
The number of participants responding to treatment, defined as a ≥ 50%, ≥ 70%, or ≥ 90% reduction from the Run-In Period in investigator-confirmed HAE attack rate (for adult participants: compared to placebo during the 6-month Treatment Period). | Baseline through Day 181
Number of participants with no investigator-confirmed HAE attacks during the 6-month Treatment Period. | Day 1 through Day 181
Change from baseline (Day 1) in the Angioedema Quality of Life questionnaire total score. | Day 1 through Day 181

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events. | Day 1 through Day 361

CONTACTS AND LOCATIONS:
Locations (79):
- United States (19):
  - Site 9, Birmingham, Alabama
  - Site 2, Scottsdale, Arizona
  - Site 3, Little Rock, Arkansas
  - Site 26, San Diego, California
  - Site 14, San Diego, California
  - Site 4, Santa Monica, California
  - Site 1, Walnut Creek, California
  - Site 8, Centennial, Colorado
  - Site 11, Colorado Springs, Colorado
  - Site 25, Tampa, Florida
  - Site 69, Weston, Florida
  - Site 43, Overland Park, Kansas
  - Site 6, Wheaton, Maryland
  - Site 67, Boston, Massachusetts
  - Site 13, Detroit, Michigan
  - Site 10, St Louis, Missouri
  - Site 7, Cincinnati, Ohio
  - Site 12, Toledo, Ohio
  - Site 15, Hummelstown, Pennsylvania
- Australia (3):
  - Site 68, Campbelltown, New South Wales
  - Site 76, Melbourne, Victoria
  - Site 74, Murdoch
- Site 45, Santo André, Brazil
- Site 28, Sofia, Bulgaria
- Canada (2):
  - Site 5, Ottawa, Ontario
  - Site 23, Edmonton
- Czechia (2):
  - Site 37, Hradec Králové
  - Site 39, Prague
- France (5):
  - Site 46, La Tronche
  - Site 54, Lille
  - Site 65, Marseille
  - Site 72, Nice
  - Site 52, Paris
- Germany (3):
  - Site 38, Berlin
  - Site 44, Frankfurt
  - Site 70, Hanover
- Site 20, Hong Kong, Hong Kong
- Site 64, Budapest, Hungary
- Israel (5):
  - Site 55, Ashkelon
  - Site 49, Haifa
  - Site 35, Petah Tikva
  - Site 34, Petah Tikva
  - Site 53, Tel Aviv
- Italy (6):
  - Site 42, Milan
  - Sie 51, Monserrato
  - Site 51, Monserrato
  - Site 66, Padua
  - Site 40, San Donato Milanese
  - Site 41, Torino
- Japan (9):
  - Site 30, Fukuoka, Kurume-shi
  - Site 56, Tsu, Mei
  - Site 61, Kawagoe, Saitama
  - Site 31, Saitama, Soka-shi
  - Site 57, Hiroshima
  - Site 50, Hiroshima
  - Site 58, Kawasaki
  - Site 47, Saga
  - Site 73, Tokyo
- Site 27, Amsterdam, Netherlands
- Site 75, Auckland, New Zealand
- Site 33, Skopje, North Macedonia
- Poland (3):
  - Site 71, Krakow
  - Site 78, Lodz
  - Site 29, Rzeszów
- Site 59, San Juan, Puerto Rico
- Site 21, Cape Town, South Africa
- South Korea (3):
  - Site 62, Seoul, Jongno
  - Site 60, Yangcheon, Seoul
  - Site 77, Seongnam-si
- Spain (4):
  - Site 32, Barcelona
  - Site 63, Madrid
  - Site 48, Seville
  - Site 36, Valencia
- United Kingdom (6):
  - Site 18, Plymouth, Devon
  - Site 24, Hampstead, London
  - Site 19, Bristol
  - Site 16, Cambridge
  - Site 22, Frimley
  - Site 17, London

IPD SHARING:
Plan to Share IPD: No